CLINICAL TRIAL: NCT06442410
Title: Comparison of Differential Target Multiplexed Spinal Cord Stimulation (DTM™ SCS) Therapy Combined With CMM to CMM Alone in the Treatment of Intractable Back Pain Subjects Without Previous History of Lumbar Surgery
Brief Title: Comparison of DTM™ SCS Therapy Combined With Conventional Medical Management (CMM) to CMM Alone in the Treatment of Intractable Back Pain Subjects Without Previous History of Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Collaborators: SGX Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MDT24011; ISRCTN10663814 (Registry Identifier: ISRCTN Registry)
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Pain, Intractable; Pain, Chronic
MeSH Terms: conditions — Pain, Intractable; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Subjects meeting study entrance criteria will be randomized in a 1:1 ratio to one of two study treatment groups:
  * DTM™ SCS programming approach with Conventional Medical Management (CMM)
  * CMM alone
  There is an optional two-way crossover to the other treatment group available for all subjects who remain in the study at the 6-months visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Group - DTM™ SCS programming approach with Conventional Medical Management (CMM) (Experimental): Subjects will undergo a Trial Phase with DTM™ SCS programming. Stimulation will be delivered from an external neurostimulator. Those who have a "successful Trial Phase" will proceed to permanent implantation of the Intellis™ SCS system to evaluate DTM™ SCS therapy and will undergo up to 24 months of stimulation delivery.
  Subjects randomized to either treatment group will have the optional possibility to crossover to the alternative treatment arm after the 6-month visit. If the subject and investigator believe that the DTM™ SCS + CMM treatment has not generated sufficient pain relief to warrant continued treatment, then the subject will be provided with the option to crossover to the CMM group. If all SCS programming attempts fail, then DTM™ SCS therapy will be switched off and the subject will continue with their CMM treatment and will visit the clinic approximately a total of 18 months follow-up in the study (i.e. 6 months DTM™ SCS and 12 months CMM).
  Interventions: Device: DTM™ spinal cord stimulation therapy delivered via Intellis™ neurostimulator system; Other: Conventional Medical Management (CMM)
- Control Group - Conventional Medical Management (CMM) alone (Active Comparator): The choice of appropriate CMM will be made by the Investigator as determined to be the best standard of care for each individual subject i.e. optimized individual conventional therapy. These treatments would be generally consistent with the American College of Physicians and the American Pain Society Guidelines as published in the Annals of Internal Medicine and European/UK guidelines. Subjects in this group will also undergo up to 24 months of CMM.
  Subjects randomized to either treatment group will have the optional possibility to crossover to the alternative treatment arm after the 6-month visit. If the subject and investigator believe that the CMM treatment has not generated sufficient pain relief to warrant continued treatment, then the subject will be provided with the option to crossover to the DTM™ SCS therapy group. Following their device activation, they will attend visits approximately a total of 18 months follow-up in the study (i.e. 6 months CMM and 12 months DTM™ SCS).
  Interventions: Other: Conventional Medical Management (CMM)

INTERVENTIONS:
Device: DTM™ spinal cord stimulation therapy delivered via Intellis™ neurostimulator system — Along with the appropriate Conventional Medical Management treatment made by the Investigator, the subject will be trialed and implanted with an Intellis™ neurostimulator system using DTM™ SCS programming parameters.
  Arms: Test Group - DTM™ SCS programming approach with Conventional Medical Management (CMM)
Other: Conventional Medical Management (CMM) — The CMM treatment can be modified at any moment by the investigators based on their clinical evaluation and local standard of care. They may also consists of one or more of the following treatments: medications, combined physical and psychological management, physical therapy, back rehabilitation program, spinal manipulation and spinal mobilization, traction, acupuncture, cognitive behavioral therapy, biofeedback, nerve blocks, radio frequency ablation, epidural steroid injections, transcutaneous electrical nerve stimulation, intradiscal electrothermal therapy, nucleoplasty, also called plasma disc decompression (PDD) or similar

SUMMARY:
The purpose of this investigational study is to document the safety, clinical effectiveness and health economic analytics of DTM™ SCS programming delivered through the Intellis™ neurostimulator in subjects with chronic, intractable pain of the trunk with or without lower limb pain, including unilateral or bilateral pain without prior history of spine surgery and refractory to conservative treatment and are not candidates for lumbar spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be a candidate for SCS system (trial and implant)
* Have been diagnosed with chronic, refractory axial low back pain with or without lower limb pain, with a neuropathic component as assessed by the investigator, 6 months refractory to conventional therapy and are not eligible for spine surgery (e.g., lumbar fusion, discectomy, laminectomy, laminotomy) at the time of enrollment
* Has an average back pain intensity ≥ 6.0 cm on the 10.0 cm Visual Analog Scale (VAS) at the time of enrollment
* Be willing and capable of giving written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the subject's participation has been provided.
* Be willing and capable of subjective evaluation, read and understand written questionnaires, and read, understand and sign the written inform consent
* Be 18 years of age or older at the time of enrollment
* Be on a stable pain medication regime, as determined by the study investigator, for at least 30 days prior to enrolling in this study
* Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

* Had a previous spinal surgery (e.g., lumbar fusion, discectomy, laminectomy, laminotomy)
* Has a medical, anatomical, and/or psychosocial condition that is contraindicated for commercially available Intellis™ SCS systems as determined by the Investigator
* Has a diagnosed back condition with inflammatory causes of back pain (e.g., onset of severe pain with activity), serious spinal pathology and/or neurological disorders as determined by the Investigator
* Be concurrently participating in another clinical study
* Has an existing active implanted device such as a pacemaker, another SCS unit, peripheral nerve stimulator, and/or drug delivery pump, etc.
* Has pain in other area(s) and/or medical condition requiring the regular use of significant pain medications that could interfere with accurate pain reporting, study procedures, and/or confound evaluation of study endpoints, as determined by the Investigator
* Has mechanical spine instability as determined by the Investigator
* Has undergone, within 30 days prior to enrollment, an interventional procedure and/or surgery to treat back and/or leg pain, which is providing significant pain relief
* Has unresolved major issues of secondary gain (e.g., social, financial, legal), as determined by the investigator
* Be involved in an injury claim under current litigation or has a pending or approved worker's compensation claim
* Be pregnant (determined by urine testing unless female subject is surgically sterile or post-menopausal. If female, sexually active, and childbearing age, subject must be willing to use a reliable form of birth control.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2023-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirit Argov, Study Director — Medtronic
Locations (12):
- Belgium (3):
  - AZ Delta, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - GZA - Sint Augustinus Ziekenhuis, Wilrijk
- Germany (2):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - München Klinik Bogenhausen, München
- Netherlands (3):
  - Rijnstate - Locatie Elst, Elst
  - Maastricht University Medical Center, Maastricht
  - Diakonessenhuis Locatie Zeist, Zeist
- Spain (4):
  - Hospital Clínico Universitario de Santiago, A Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ISRCTN Registry posting — https://doi.org/10.1186/ISRCTN10663814

RESULTS

PARTICIPANT FLOW:
Period: Overall Non-Crossover
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Started | 55 | 57
Completed (50 subjects in Control Group crossed over to Test Group at 6-month optional crossover timepoint. No Test Group subject crossed over to Control Group at 6-month optional crossover time point.) | 40 | 4
Not Completed | 15 | 53
Period: Optional Crossover at 6 Month
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Started | 0 | 50 (No Test Group subject crossed over to Control Group at 6 month optional crossover timepoint.)
Completed | 0 | 39 (No Test Group subject crossed over to Control Group at 6 month optional crossover timepoint.)
Not Completed | 0 | 11

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included Modified Intent to Treat (mITT) population, defined as all successfully randomized subjects to the test arm who completed the Trial Phase and all successfully randomized subjects to the control arm.
Groups:
- Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM): Subjects will undergo a Trial Phase with DTM™ SCS programming. Stimulation will be delivered from an external neurostimulator. Those who have a "successful Trial Phase" will proceed to permanent implantation of the Intellis™ SCS system to evaluate DTM™ SCS therapy and will undergo up to 24 months of stimulation delivery.
  Subjects randomized to either treatment group will have the optional possibility to crossover to the alternative treatment arm after the 6-month visit. If the subject and investigator believe that the DTM™ SCS + CMM treatment has not generated sufficient pain relief to warrant continued treatment, then the subject will be provided with the option to crossover to the CMM group. If all SCS programming attempts fail, then DTM™ SCS therapy will be switched off and the subject will continue with their CMM treatment and will visit the clinic approximately a total of 18 months follow-up in the study (i.e. 6 months DTM™ SCS and 12 months CMM).
  DTM™ spinal cord stimulation therapy delivered via Intellis™ neurostimulator system: Along with the appropriate Conventional Medical Management treatment made by the Investigator, the subject will be trialed and implanted with an Intellis™ neurostimulator system using DTM™ SCS programming parameters.
- Total: Total of all reporting groups
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone | Total
Number analyzed (Participants) | 51 | 57 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.86 (13.01) | 56.86 (12.81) | 56.39 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 22 | 29 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 14 | 16 | 30
  Belgium | 18 | 23 | 41
  Germany | 3 | 3 | 6
  Spain | 16 | 15 | 31
Years with Chronic Low Back Pain (CLBP), Continuous [Mean (Standard Deviation); unit: years] | 10.4 (10.9) | 11.6 (10.8) | 11.0 (10.8)
Body Mass Index (BMI), Continuous [Mean (Standard Deviation); unit: kg/m²] | 27.54 (4.50) | 27.81 (4.42) | 27.68 (4.44)
Baseline Back Pain Visual Analog Scale (VAS), Continuous [Mean (Standard Deviation); unit: cm] — Visual Analog Scale is a scaled psychometric instrument to report pain severity on a 10 cm line, with 0 indicating no pain and 10 indicating the worst pain imaginable.
  cm | 7.91 (0.97) | 7.76 (1.03) | 7.83 (1.00)
Pain Diagnosis [Count of Participants; unit: Participants]
  Chronic intractable back pain | 51 | 57 | 108
  Chronic intractable leg pain | 43 | 50 | 93

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Individual Responders
Description: Individual Responders defined as decrease in back pain rating on 10 cm Visual Analog Scale (VAS) by at least 50%. Visual Analog Scale is a scaled psychometric instrument to report pain severity on a 10 cm line, with 0 indicating no pain and 10 indicating the worst pain imaginable.
Time Frame: 6 months
Population: Modified Intent to Treat (mITT): All successfully randomized subjects to the test arm who completed the Trial Phase and all successfully randomized subjects to the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 47 | 56
Participants | 40 | 2
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

2. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 1 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 49 | 57
Participants | 41 | 1
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

3. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 48 | 56
Participants | 41 | 3
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

4. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 9 months
Population: Modified Intent to Treat (mITT): All successfully randomized subjects to the test arm who completed the Trial Phase and all successfully randomized subjects to the control arm. Crossover subjects were counted as failures (i.e. non-responders) for endpoints defined in terms of responders in their group of original randomization assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 56
Participants | 37 | 0
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

5. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 55
Participants | 36 | 0
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

6. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 18 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 55
Participants | 37 | 1
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Superiority; p < 0.0001, Chi-squared

7. Secondary Outcome: Percentage of Individual Responders
Description: as for outcome 1
Time Frame: 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 43 | 55
Participants | 38 | 3

8. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: Change from Baseline in Back Pain 10 cm VAS = Follow-up Visit Pain VAS - Baseline Pain VAS. A negative result reflects a decrease in the Pain VAS, while a positive result reflects an increase in Pain VAS. Visual Analog Scale is a scaled psychometric instrument to report pain severity on a 10 cm line, with 0 indicating no pain and 10 indicating the worst pain imaginable.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 49 | 57
cm | -5.69 (2.17) | -0.36 (1.46)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

9. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 48 | 56
cm | -5.77 (2.04) | -0.40 (1.74)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

10. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 47 | 56
cm | -5.76 (2.07) | 0.13 (1.55)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

11. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 9 months
Population: Modified Intent to Treat (mITT): All successfully randomized subjects to the test arm who completed the Trial Phase and all successfully randomized subjects to the control arm. Crossover subjects were counted as failures (i.e. non-responders) for endpoints defined in terms of responders in their group of original randomization assignment, carrying forward the baseline (pre-treatment) scores.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 56
cm | -5.43 (2.13) | -0.07 (0.59)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

12. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 55
cm | -5.42 (2.23) | -0.10 (0.42)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

13. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 18 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 45 | 55
cm | -5.52 (1.93) | -0.16 (0.73)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

14. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Back Pain Score
Description: as for outcome 8
Time Frame: 24 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone
Number analyzed (Participants) | 43 | 55
cm | -5.98 (1.68) | -0.22 (0.95)
Statistical Analysis 1: Comparison: Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) vs Control Group - Conventional Medical Management (CMM) Alone; Test type: Non-Inferiority — A non-inferiority margin of 0.65 cm was selected based on a previous study of a similar therapy against traditional SCS; p < 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: From enrollment through the completion of the study (up to 24 months follow-up)
Description: Adverse events were captured from enrollment through the completion of the study (up to 24 months follow-up).
  As the primary efficacy measure in this study is pain, back or leg pain does not need to be reported as an adverse event unless it meets the definition of a serious adverse event. However, Investigators may, at their discretion, report any pain-related adverse events during the study.
Groups:
- Optional Crossover at 6 Month: Subjects randomized to either treatment group will have the optional possibility to crossover to the alternative treatment arm after the 6-month visit.
Arm/Group | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) | Control Group - Conventional Medical Management (CMM) Alone | Optional Crossover at 6 Month
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/57 | 0/50
Serious Adverse Events (participants affected / at risk) | 15/55 | 3/57 | 10/50
Other Adverse Events (participants affected / at risk) | 29/55 | 6/57 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) (N=55) | Control Group - Conventional Medical Management (CMM) Alone (N=57) | Optional Crossover at 6 Month (N=50)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Drug-induced liver inquiry (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adhesiolysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group - DTM™ SCS Programming Approach With Conventional Medical Management (CMM) (N=55) | Control Group - Conventional Medical Management (CMM) Alone (N=57) | Optional Crossover at 6 Month (N=50)
COVID-19 (Infections and infestations) | 14 (14) | 3 (3) | 14 (14)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 3 (3) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT06442410/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT06442410/SAP_001.pdf